CLINICAL TRIAL: NCT05094596
Title: ATATURK UNİVERSITY
Brief Title: Effect of Montelukast Therapy on Clinical Course, Pulmonary Function, and Mortality in Patients With COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bugra Kerget (Other)
Responsible Party: Sponsor-Investigator, Bugra Kerget, Associate professor, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATATURK-BUGRA-001
Record Dates: First submitted 2021-10-21; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — montelukast; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standart treatment group (Experimental): Standard treatment in accordance with our national COVID-19 diagnosis and treatment guide
  Interventions: Drug: Standart treatment group
- Montelukast sodium 10 mg treatment (Experimental): Received 10 mg/day oral montelukast in addition to standard treatment
  Interventions: Drug: Standart treatment group; Drug: Montelukast sodium 10 mg treatment
- Montelukast sodium 20 mg treatment (Experimental): Received 10 mg/day oral montelukast in addition to standard treatment
  Interventions: Drug: Standart treatment group; Drug: Montelukast sodium 20 mg treatment

INTERVENTIONS:
Drug: Standart treatment group — Group 1 (n=60) received standard treatment in accordance with our national COVID-19 diagnosis and treatment guide.
Drug: Montelukast sodium 10 mg treatment — Group 2 (n=60) received 10 mg/day oral montelukast in addition to standard treatment
  Arms: Montelukast sodium 10 mg treatment
Drug: Montelukast sodium 20 mg treatment — Group 3 (n=60) were given 20 mg/day oral montelukast in addition to standard treatment.
  Arms: Montelukast sodium 20 mg treatment

SUMMARY:
'Pandemic' is a medical term that has become a ubiquitous part of the global vocabulary over the last year. Although pandemics have occurred throughout human history, their sociocultural, economic, and psychological impact can leave lasting damage. In the current COVID-19 pandemic, more than 200 million confirmed cases of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection have been reported to date. While most people present with mild symptoms such as loss of taste and smell, sore throat, joint pain, and headache, it can cause serious morbidity and mortality, especially in individuals over 65 years of age and those with comorbidities .

Acute respiratory distress syndrome (ARDS) and macrophage activation syndrome (MAS) are among the main causes of morbidity and mortality in COVID-19. A contributing factor in the development of these clinical conditions is overproduction of proinflammatory cytokines, primarily tumor necrosis factor alpha (TNF-α), interleukin-6 (IL-6), IL-8, and IL-1β. These cytokines cause increased leukocyte accumulation in the alveolar spaces and consequently an increase in reactive oxygen radicals and proteases, which inevitably leads to capillary endothelial damage and alveolar epithelial damage .

Montelukast is a potent cysteinyl leukotriene (cysLT) receptor antagonist with anti-inflammatory activity and has been proven to significantly suppress oxidative stress. Moreover, cysLTs also have an important role in the regulation of cytokine production. Administration of high doses of montelukast reduces IL-4, IL-5, and IL-13 production by T helper 2 cells . This effect makes it an important anti-inflammatory agent in the treatment of asthma. In addition, montelukast was shown to significantly inhibit bradykinin-induced tracheal smooth muscle contraction, thus supporting an interaction between bradykinin and leukotriene mediators .

In studies investigating the efficacy of cysLT for ARDS and MAS, montelukast was found to increase interferon gamma (IFN-γ) production and significant decrease the production of proinflammatory cytokines such as IL-1β, IL-6, and IL-8 in mice infected with respiratory syncytial virus. In another study, cysLT prevented neutrophil infiltration, lung inflammation, and oxidative stress and significantly decreased levels of TNF-α and IL-6 in both the lung parenchyma and bronchoalveolar lavage fluid in an animal model of ARDS induced by hemorrhagic shock.

In this study, the investigators aimed to investigate the effect of treatment with varying doses of montelukast as an adjunct to standard antiviral therapy on pulmonary function tests and clinical course in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* The prospective controlled randomized study included patients who presented to the emergency department of Erzurum Regional Training and Research Hospital with history of travel abroad within the last 14 days or contact with a confirmed or suspected COVID-19 patient and had recent complaints of fever, cough, dyspnea, malaise, and sudden loss of taste and smell. Patients regarded as high risk for COVID-19 underwent standard high-resolution computed tomography (HRCT). Predominantly peripheral bilateral ground glass opacities, subsegmental consolidation or linear opacities, crazy-paving pattern, and reverse halo sign were considered typical HRCT findings for COVID-19. Patients with these findings and patients with radiologically atypical findings but consistent clinical symptoms were hospitalized with suspected COVID-19. The diagnosis was confirmed by SARS-CoV-2 real-time polymerase chain reaction (PCR) testing of nasopharyngeal swab samples.

Exclusion Criteria:

* Patients with any potential contraindications to pulmonary function testing (recent myocardial infarction, pulmonary embolism, cerebral aneurysm, active hemoptysis, pneumothorax, nausea/vomiting, recent thoracic, abdominal, or ocular surgery) were excluded before testing. In addition, patients who developed ARDS or MAS associated with secondary bacterial infection during the first week of treatment were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-10-22 (Estimated); Primary Completion 2021-12-22 (Estimated); Study Completion 2022-01-22 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test | 3 month
  Pulmonary function tests were performed in a negative-pressure room by a technician wearing protective equipment to prevent transmission. Before testing, patients were instructed to abstain from smoking (24 hours), alcohol (4 hours), strenuous exercise (30 minutes), and heavy meals (2 hours). The patients' age, height, and weight were recorded. Tests were performed with the patients lightly dressed and BTPS correction was performed according to room air and barometric pressure. The technician explained the maneuver to the patients and three acceptable spirograms were obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No